CLINICAL TRIAL: NCT04827654
Title: The Impact of Providing Choices for Fruits and Vegetable Access on Child Diet
Brief Title: Increasing Adoption of Fruits and Vegetables Into Family Diet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Collaborators: Boys and Girls Club of Austin (Unknown)
Responsible Party: Principal Investigator, Maninder Kahlon, Associate Professor, University of Texas at Austin
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 00000566
Record Dates: First submitted 2021-03-29; First posted 2021-04-01 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Diet, Healthy

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial, outcomes on reference child and reference caregiver; In the intervention arm, fruits and vegetables and vouchers cover more than 1 cup a day increase for families, using an average of 5 people as family size.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Individuals collecting data will be blinded to the participant randomization status.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Families in the intervention arm will receive a program of 4 weeks of access to fruit and vegetables through direct access (produce box) and a gift card to the grocery store for purchase of preferred produce.
  Interventions: Dietary Supplement: Weekly produce box and gift card
- Control Group (No Intervention): Families in the control group will not receive any produce boxes or gift cards during the study period. At the end of the study period they will receive gift cards of equivalent amount.

INTERVENTIONS:
Dietary Supplement: Weekly produce box and gift card — Weekly box of produce (5-10 lbs) and $10.00 gift card to a local grocery store to purchase preferred produce. If progress on self-goals completed, an additional $10.00 card provided, weekly, for 3 weeks.
  Arms: Intervention group

SUMMARY:
The investigators are interested in maximizing the consumption of fruits and vegetables (F&V) in elementary school children by increasing the access to F&V by providing them in the home environment via direct delivery (F&V bag & recipes) and a gift card to purchase preferred choices. This also decreases barriers to trying F&V and switching to a more F&V-focused diet, e.g., access, cost, knowledge of what to do with fruits and vegetables by their families in household diet, and a period of time to try and get used to more F&V in the diet without worrying about access and cost.

We hypothesize that at the end of 4 weeks, children in families that were given access to a F&V produce box with associated recipes, a gift card to purchase preferred choices, and a cooking incentive kit, consumed significantly better diets as measured with a diet composite score compared with children in families who did not receive increased F&V access.

ELIGIBILITY:
Inclusion Criteria:

1. Families must be participants in the Boys and Girls "Club on the Go" program. They could sign up to become a participant while we are recruiting.
2. Caregiver must be able to come to the same "Club on the Go" site every week.
3. At least one child in the family must be k-5 student.
4. Caregiver must be able to read and write in English or Spanish to answer assessments.

Exclusion Criteria:

1. Reference child with any medical condition in which they have to follow a specific diet.
2. Caregiver cannot read and write in English or Spanish.
3. Reference child not living with caregiver for majority of time (75% or greater).
4. Families that do not meet the inclusion criteria

Ages: 4 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 68 (Actual)
Dates: Start 2021-03-31 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
School Physical Activity and Nutrition (SPAN) questionnaire elementary version | 24 hours
  dietary recall measure for fruit and vegetables scale of 0-12 with higher scores equating to more vegetable consumption

CONTACTS AND LOCATIONS:
Overall Officials: Maninder Kahlon, PhD, Principal Investigator — University of Texas at Austin
Locations (7):
- United States (7):
  - Booker T. Washington, Austin, Texas
  - Chalmers Court, Austin, Texas
  - Meadowbrook Elementary School, Austin, Texas
  - Home Club, Austin, Texas
  - Walnut Creek Elementary School, Austin, Texas
  - NYOS Kramer, Austin, Texas
  - Elgin High School, Elgin, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Olsho LE, Klerman JA, Wilde PE, Bartlett S. Financial incentives increase fruit and vegetable intake among Supplemental Nutrition Assistance Program participants: a randomized controlled trial of the USDA Healthy Incentives Pilot. Am J Clin Nutr. 2016 Aug;104(2):423-35. doi: 10.3945/ajcn.115.129320. Epub 2016 Jun 22. PMID 27334234
- [Result] Sharma SV, Markham C, Chow J, Ranjit N, Pomeroy M, Raber M. Evaluating a school-based fruit and vegetable co-op in low-income children: A quasi-experimental study. Prev Med. 2016 Oct;91:8-17. doi: 10.1016/j.ypmed.2016.07.022. Epub 2016 Jul 25. PMID 27471022
- [Result] Seligman HK, Smith M, Rosenmoss S, Marshall MB, Waxman E. Comprehensive Diabetes Self-Management Support From Food Banks: A Randomized Controlled Trial. Am J Public Health. 2018 Sep;108(9):1227-1234. doi: 10.2105/AJPH.2018.304528. Epub 2018 Jul 19. PMID 30024798
- [Derived] Kahlon MK, Aksan NS, Aubrey R, Barnes J, Clark N, Cowley-Morillo M, Engelman L, Guerra J, Guevara A, Marshall A, Hoelscher DM. Effect of Brief Produce Exposure and Unconstrained Grocery Gift Cards on Caregiver Influence on Diet of Elementary Age Children: A Randomized Clinical Trial. JAMA Netw Open. 2022 May 2;5(5):e2212973. doi: 10.1001/jamanetworkopen.2022.12973. PMID 35622367